CLINICAL TRIAL: NCT03848091
Title: Prosthesis Infection and One-step Exchange: Pretreatment by Targeted Antibiotic Therapy in
Brief Title: Prosthesis Infection and One-step Exchange: Pretreatment by Targeted Antibiotic Therapy in At-risk Patients
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, CRA, Hospices Civils de Lyon
Other Study IDs: 18-030
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prosthetic Joint Infection; Antibiotic Resistant Infection
Keywords: bone and joint infection; Antibiotic pretreatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antibiotic pretreatment: patients having had an antibiotic pretreatment before a one-step exchange arthroplasty
  Interventions: Other: Antibiotic pretreatment

INTERVENTIONS:
Other: Antibiotic pretreatment — a strategy with antibiotic pretreatment before one-step exchange arthroplasty in patients who bacteria responsible for the infection has been indentified (puncture, blood cultures,...)

SUMMARY:
One-step exchange arthroplasty is more and more used in the treatment of chronic infections, especially in patients at risk anesthetic.

This strategy is not recommended in patients infected with multidrug-resistant organisms or difficult to treat because of a risk of bacterial persistence on the new implant.

Antibiotic pretreatment by a narrow-spectrum molecule and for which resistance acquisition is difficult might be of interest to try to reduce the inoculum and avoid contamination of the new implant.

ELIGIBILITY:
Inclusion Criteria:

* patients having had a antibiotic pretreatment targeted before a one step exchange arthroplasty

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having had a antibiotic pretreatment targeted before a one step exchange arthroplasty managed at the Croix-Rousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

SECONDARY OUTCOMES:
rate of use of this strategy | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  descriptions of patients managed with this strategy
rate of bacteria responsible for infection | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  bacterial epidemiology

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Md,PhD, Principal Investigator — HCL
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided